CLINICAL TRIAL: NCT04916002
Title: A Multicenter, Open-label, Phase 2 Study of Intratumoral Vidutolimod (CMP-001) in Combination With Intravenous Cemiplimab in Subjects With Selected Types of Advanced or Metastatic Cancer
Brief Title: A Trial To Find Out If Vidutolimod Together With Cemiplimab Is Safe And If It Works In Adult Participants With Advanced Cancer Or Metastatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision related to study drug supply
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMP-001-009; 2023-507344-36-01 (Registry Identifier: EUCT Number)
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Merkel Cell Carcinoma; Cutaneous Squamous Cell Carcinoma; Basal Cell Carcinoma; Triple Negative Breast Cancer; Non-Small Cell Lung Cancer; Oropharynx Squamous Cell Carcinoma
Keywords: vidutolimod; Metastatic Cancer; Advanced Cancer; MCC; CSCC; BCC; TNBC; NSCLC; OPSCC
MeSH Terms: conditions — Carcinoma, Merkel Cell; Carcinoma, Basal Cell; Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Vidutolimod and cemiplimab for cutaneous squamous cell carcinoma (CSCC) (A1) (Experimental): Participants who have not received prior systemic therapy for metastatic or locally and/or regionally advanced unresectable CSCC and who are not eligible for curative radiation will receive vidutolimod intratumoral(ly) (IT) and cemiplimab intravenous (IV) according to the treatment schedule until a reason for treatment discontinuation is reached.
  Interventions: Drug: vidutolimod; Drug: cemiplimab
- Vidutolimod and cemiplimab for CSCC (A2) (Experimental): Participants who have progressed while receiving a programmed cell death protein 1 (PD-1)-blocking antibody or within 12 weeks of discontinuation of PD-1 blocking antibody for metastatic or locally and/or regionally advanced unresectable CSCC, will receive vidutolimod IT and cemiplimab IV according to the treatment schedule until a reason for treatment discontinuation is reached.
  Interventions: Drug: vidutolimod; Drug: cemiplimab
- Vidutolimod and cemiplimab for Merkel cell carcinoma (MCC) (B1) (Experimental): Participants who have not received prior systemic therapy for metastatic or locally and/or regionally advanced unresectable MCC will receive vidutolimod IT and cemiplimab IV according to the treatment schedule until a reason for treatment discontinuation is reached.
  Interventions: Drug: vidutolimod; Drug: cemiplimab
- Vidutolimod and cemiplimab for MCC (B2) (Experimental): Participants who have progressed while receiving a PD-1-blocking antibody or within 12 weeks of discontinuation of the PD-1 blocking antibody, will receive vidutolimod IT and cemiplimab IV according to the treatment schedule until a reason for treatment discontinuation is reached.
  Interventions: Drug: vidutolimod; Drug: cemiplimab
- Vidutolimod and cemiplimab for triple negative breast cancer (TNBC) (C1) (Experimental): Participants who have not received prior therapy with immune checkpoint inhibitors (iCPIs) and who must have previously received treatment with sacituzumab govitecan (all advanced or metastatic TNBC participants), with trastuzumab deruxtecan [human epidermal growth factor receptor 2 (HER2)-low participants] and with adenosine diphosphate ribose polymerase (PARP) inhibitor [for BReast CAncer gene (BRCA)] for TNBC will receive vidutolimod IT and cemiplimab IV according to the treatment schedule until a reason for treatment discontinuation is reached.
  Interventions: Drug: vidutolimod; Drug: cemiplimab
- Vidutolimod and cemiplimab for TNBC (C2) (Experimental): Participants who have previously received treatment with sacituzumab govitecan (all advanced or metastatic TNBC participants), with trastuzumab deruxtecan (HER2-low participants) and with PARP inhibitor (for BRCA) and who have progressed while receiving a PD-1-blocking antibody or within 12 weeks of discontinuation of a PD-1 blocking antibody for advanced or metastatic TNBC, will receive vidutolimod IT and cemiplimab IV according to the treatment schedule until a reason for treatment discontinuation is reached.
  Interventions: Drug: vidutolimod; Drug: cemiplimab
- Vidutolimod and cemiplimab for basal cell carcinoma (BCC) (D) (Experimental): Participants who have not received prior hedgehog pathway inhibitor therapy, or prior anti-PD-1/programmed cell death ligand 1 (PD-L1) therapy and who do not wish to receive or who are not candidates for a hedgehog inhibitor, for metastatic or locally and/or regionally advanced unresectable BCC and will receive vidutolimod IT and cemiplimab IV according to the treatment schedule until a reason for treatment discontinuation is reached.
  Interventions: Drug: vidutolimod; Drug: cemiplimab
- Vidutolimod and cemiplimab for non-small cell lung cancer (NSCLC) (E) (Experimental): Participants with advanced NSCLC (locally advanced who are not candidates for surgical resection or definitive chemoradiation or metastatic) whose tumors have high PD-L1 expression [tumor proportion score (TPS) ≥50%] based on a prior PD-L1 result as determined by College of American Pathologists (CAP)/Clinical Laboratory Improvement Amendments (CLIA) (or equivalently licensed) lab, with no epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK) or ros oncogene 1 (ROS1) aberrations, and who have not received prior anti-PD-1/PD-L1 therapy and are amenable to IT therapy and do not wish to receive chemotherapy.
  Note: this cohort is not conducted in Europe
  Interventions: Drug: vidutolimod; Drug: cemiplimab
- Vidutolimod and cemiplimab for recurrent/metastatic Oropharynx Squamous Cell Carcinoma (OPSCC) (F) (Experimental): Participants with PD-L1 combined positive score (CPS) ≥ 1, based on a prior PD-L1 result and human papillomavirus (HPV)-positive disease based on a prior result, who have not received prior systemic therapy for recurrent/metastatic disease. Participants will receive vidutolimod IT and cemiplimab IV according to the treatment schedule until a reason for treatment discontinuation is reached.
  Interventions: Drug: vidutolimod; Drug: cemiplimab

INTERVENTIONS:
Drug: vidutolimod — Participants will receive vidutolimod for up to 2 years as follows: 10 mg IT weekly for 7 doses after which vidutolimod will be administered every 3 weeks (Q3W). The first dose of vidutolimod may be administered subcutaneously (SC) or IT at the discretion of Investigator. All subsequent doses will be IT. The initial 7 doses of vidutolimod, delivered on a weekly dosing schedule, must be completed before starting the Q3W vidutolimod dosing schedule.
  Other Names: CMP-001
Drug: cemiplimab — Participants will receive cemiplimab for up to 2 years as follows: 350 mg IV infusion over 30 minutes at week 1 dose 1 (W1D1) and Q3W thereafter.
  Other Names: Libtayo; REGN2810

SUMMARY:
The goal of this study is to learn if giving cemiplimab and vidutolimod together could be effective in treating advanced cancer. The main questions it aims to answer are:

* How many participants' cancers respond to vidutolimod together with cemiplimab?
* Is vidutolimod together with cemiplimab safe and well-tolerated?
* How well does vidutolimod together with cemiplimab treat participants' cancer?

Participants will receive trial treatment for up to 2 years. 30 days after stopping treatment, participants will have a follow-up visit. After that visit, the trial staff will continue to follow up with participants about every 3 months, until the trial ends.

DETAILED DESCRIPTION:
Former Sponsor Checkmate Pharmaceuticals Note: Early termination planned on 31Oct2024 due to study drug supply

ELIGIBILITY:
Key Inclusion Criteria:

Participants enrolled in the study must meet all of the following inclusion criteria to be eligible.

1. Histopathologically-confirmed diagnosis of cancer, as defined by the protocol.
2. Measurable disease, as defined by RECIST v1.1 and as defined in the protocol. Note: CSCC, MCC and BCC subjects without radiographically measurable disease are not excluded if there is at least 1 lesion ≥ 10 mm in at east 1 dimension documented by color photography.
3. Adequate organ function based on most recent laboratory values within 3 weeks before first dose of study treatment on Week 1 Day 1 (W1D1), as defined in the protocol.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1 at Screening.

Key Exclusion Criteria:

Participants presenting with any of the following will not qualify for entry into the study:

1. Received radiation therapy (or other non-systemic therapy) within 2 weeks before first dose of study treatment on W1D1. Participants should have recovered (i.e. Grade ≤ 1 or at baseline) from radiation-related toxicities.
2. Had major surgeries (including complete oncologic resection) within last 4 weeks prior to enrollment, and/or have not recovered adequately from the toxicities and/or complications from the intervention. Minor surgeries (including routine resections of early stage CSCCs and BCCs that may be due to field cancerization) require a 7-day washout.
3. Received systemic pharmacologic doses of corticosteroids > 10 mg/day prednisone within 15 days before first dose of study treatment on W1D1, as defined in the protocol.
4. History of immune-mediated AE leading to permanent discontinuation due to prior PD-1-blocking antibody.
5. Not fully recovered from AEs due to prior treatment (to Grade 1 or less, per Common Terminology Criteria for Adverse Events (CTCAE), with the exception of persistent vitiligo, alopecia, hypothyroidism, diabetes mellitus, and adrenal and/or pituitary insufficiency.
6. Active pneumonitis or history of noninfectious pneumonitis that required steroids.
7. Severe uncontrolled medical disease within 12 months of screening, including but not limited to poorly controlled hypertension, unstable angina, myocardial infarction, congestive heart failure (New York Heart Association Class II or greater), pericarditis, cerebrovascular accident, or implanted or continuous use of a pacemaker or defibrillator, or emphysema with FEV1 ≤ 50% predicted.
8. Known history of immunodeficiency.
9. Known additional malignancy that is progressing or required active treatment within the past 3 years, as defined in the protocol.
10. Active autoimmune disease that required systemic treatment in past 2 years; replacement therapy is not considered a form of systemic treatment.
11. Untreated, symptomatic, or enlarging central nervous system metastases or carcinomatous meningitis (including leptomeningeal metastases from solid tumors).

NOTE: Other protocol defined Inclusion/Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (24):
- United States (20):
  - University of Alabama, Birmingham, Alabama
  - City of Hope, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California, Los Angeles, California
  - GenesisCare USA, Jacksonville, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - University of Iowa, Iowa City, Iowa
  - Norton Cancer Institute, Louisville, Kentucky
  - VA Maryland Health Care System, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Dartmouth Clinical Trial Office, Lebanon, New Hampshire
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - East Carolina University, Greenville, North Carolina
  - Ohio State University, Columbus, Ohio
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Oncology Consultants, Houston, Texas
  - University of Utah Huntsman Cancer Center, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
- Australia (4):
  - St. Vincent's Hospital, Darlinghurst, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Peter MacCallum Cancer Centre (PMCC) and The Royal Melbourne Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A1: CMP-001+Cemiplimab for CSCC: Participants who have not received prior systemic therapy for advanced cutaneous squamous cell carcinoma (CSCC) received CMP-001 intratumorally (IT) + cemiplimab intravenously (IV) according to the treatment schedule
- Cohort A2: CMP-001+Cemiplimab for CSCC: Participants who have progressed on prior programmed cell death protein 1 (PD-1) therapy for advanced CSCC received CMP-001 IT + cemiplimab IV according to the treatment schedule
- Cohort B1: CMP-001+Cemiplimab for MCC: Participants who had not received prior systemic therapy for advanced merkel cell carcinoma (MCC) received CMP-001 IT + cemiplimab IV according to the treatment schedule
- Cohort B2: CMP-001+Cemiplimab for MCC: Participants who have progressed on prior PD-1 therapy for advanced MCC received CMP-001 IT + cemiplimab IV according to the treatment schedule
- Cohort D: CMP-001+Cemiplimab for BCC: Participants who have not received prior systemic therapy for advanced BCC (hedgehog pathway inhibitor or anti-PD-1/programmed cell death ligand 1 [PD-L1]) received CMP-001 IT + cemiplimab IV according to the treatment schedule
Period: Overall Study
Arm/Group | Cohort A1: CMP-001+Cemiplimab for CSCC | Cohort A2: CMP-001+Cemiplimab for CSCC | Cohort B1: CMP-001+Cemiplimab for MCC | Cohort B2: CMP-001+Cemiplimab for MCC | Cohort D: CMP-001+Cemiplimab for BCC
Started | 25 | 19 | 13 | 16 | 4
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 25 | 19 | 13 | 16 | 4
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 1 | 0
Not completed — Death | 8 | 7 | 4 | 9 | 0
Not completed — Study Terminated by Sponsor | 11 | 10 | 8 | 5 | 4
Not completed — End of trial | 1 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 1 | 0 | 0
Not completed — Participant non-compliance | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A1: CMP-001+Cemiplimab for CSCC | Cohort A2: CMP-001+Cemiplimab for CSCC | Cohort B1: CMP-001+Cemiplimab for MCC | Cohort B2: CMP-001+Cemiplimab for MCC | Cohort D: CMP-001+Cemiplimab for BCC | Total
Number analyzed (Participants) | 25 | 19 | 13 | 16 | 4 | 77
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.5 (14.09) | 67.9 (9.42) | 71.0 (11.55) | 69.2 (13.20) | 54.5 (9.40) | 68.8 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 5 | 5 | 0 | 23
  Male | 19 | 12 | 8 | 11 | 4 | 54
Race/Ethnicity, Customized [Number; unit: Participants] — Race Customized
  Participants
    White | 22 | 15 | 12 | 15 | 4 | 68
    Black or African American | 0 | 1 | 0 | 0 | 0 | 1
    Asian | 1 | 0 | 0 | 0 | 0 | 1
    American Indian / Alaskan Native | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Not Reported | 0 | 1 | 1 | 0 | 0 | 2
    Other | 2 | 2 | 0 | 1 | 0 | 5
Race/Ethnicity, Customized [Number; unit: Participants] — Ethnicity Customized
  Participants
    Hispanic or Latino | 4 | 0 | 1 | 1 | 0 | 6
    Not Hispanic or Latino | 21 | 18 | 12 | 15 | 4 | 70
    Not Reported | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the Percent of participants with a confirmed objective response of complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) by investigator assessment
Time Frame: Up to 31.5 Months
Population: Full Analysis Set (FAS) includes all enrolled participants who received any study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A1: CMP-001+Cemiplimab for CSCC | Cohort A2: CMP-001+Cemiplimab for CSCC | Cohort B1: CMP-001+Cemiplimab for MCC | Cohort B2: CMP-001+Cemiplimab for MCC | Cohort D: CMP-001+Cemiplimab for BCC
Number analyzed (Participants) | 25 | 19 | 13 | 16 | 4
Percentage of participants | 44.0 [24.4 to 65.1] | 5.3 [0.1 to 26.0] | 46.2 [19.2 to 74.9] | 6.3 [0.2 to 30.2] | 25.0 [0.6 to 80.6]

2. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE), Any Serious TEAE, and Any TEAE Leading to Discontinuation or Death
Description: Number of participants with any treatment-emergent adverse event (TEAE), any serious TEAE, and any TEAE leading to discontinuation or death reported.
Time Frame: Up to 31.5 months
Population: Safety Analysis Set (SAF) included all enrolled participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: CMP-001+Cemiplimab for CSCC | Cohort A2: CMP-001+Cemiplimab for CSCC | Cohort B1: CMP-001+Cemiplimab for MCC | Cohort B2: CMP-001+Cemiplimab for MCC | Cohort D: CMP-001+Cemiplimab for BCC
Number analyzed (Participants) | 25 | 19 | 13 | 16 | 4
Participants
  Any TEAE | 25 | 19 | 13 | 16 | 4
  Any serious TEAE | 14 | 10 | 6 | 11 | 2
  Any TEAE leading to discontinuation | 5 | 4 | 3 | 4 | 0
  Any TEAE leading to death | 4 | 0 | 0 | 1 | 0

3. Secondary Outcome: Severity of TEAEs as Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
Description: Number of participants per NCI CTCAE version 5.0 Adverse Event Grade reported:
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated Grade 2 Moderate; minimal, local, or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily living Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limited self-care activities of daily living Grade 4 Life-threatening consequences: urgent intervention indicated Grade 5 Death related to adverse event
Time Frame: Up to 31.5 months
Population: Safety Analysis Set (SAF) included all enrolled participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: CMP-001+Cemiplimab for CSCC | Cohort A2: CMP-001+Cemiplimab for CSCC | Cohort B1: CMP-001+Cemiplimab for MCC | Cohort B2: CMP-001+Cemiplimab for MCC | Cohort D: CMP-001+Cemiplimab for BCC
Number analyzed (Participants) | 25 | 19 | 13 | 16 | 4
Participants
  Grade 1 Mild | 2 | 2 | 2 | 2 | 0
  Grade 2 Moderate | 6 | 6 | 6 | 4 | 1
  Grade 3 Severe | 11 | 10 | 2 | 8 | 3
  Grade 4 Life-threatening | 1 | 1 | 3 | 1 | 0
  Grade 5 Death | 4 | 0 | 0 | 1 | 0
  Missing | 1 | 0 | 0 | 0 | 0

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from date of first documented response (CR or PR) to date of documented progressive disease (PD), based on RECIST v1.1, per investigator
Time Frame: Up to 31.5 months
Population: Number of participants analyzed for DOR included only participants with confirmed complete response (CR) or partial response (PR)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A1: CMP-001+Cemiplimab for CSCC | Cohort A2: CMP-001+Cemiplimab for CSCC | Cohort B1: CMP-001+Cemiplimab for MCC | Cohort B2: CMP-001+Cemiplimab for MCC | Cohort D: CMP-001+Cemiplimab for BCC
Number analyzed (Participants) | 11 | 1 | 6 | 1 | 1
Months | 11.3 [3.5 to NA] — Insufficient number of participants with events for estimated upper confidence interval | NA [NA to NA] — Median duration of DOR not reached; Insufficient number of participants with events for estimated lower and upper confidence interval | NA [4.2 to NA] — Median duration of DOR not reached; Insufficient number of participants with events for estimated upper confidence interval | NA [NA to NA] — Median duration of DOR not reached; Insufficient number of participants with events for estimated lower and upper confidence interval | NA [NA to NA] — Median duration of DOR not reached; Insufficient number of participants with events for estimated lower and upper confidence interval

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from date of first dose of study treatment to date of documented PD based on RECIST v1.1 or death, whichever occurs first
Time Frame: Up to 31.5 months
Population: Full Analysis Set (FAS) includes all enrolled participants who received any study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A1: CMP-001+Cemiplimab for CSCC | Cohort A2: CMP-001+Cemiplimab for CSCC | Cohort B1: CMP-001+Cemiplimab for MCC | Cohort B2: CMP-001+Cemiplimab for MCC | Cohort D: CMP-001+Cemiplimab for BCC
Number analyzed (Participants) | 25 | 19 | 13 | 16 | 4
Months | 10.3 [5.6 to NA] — Insufficient number of participants with events for estimated upper confidence interval | 2.0 [1.5 to 3.9] | 10.4 [4.0 to NA] — Insufficient number of participants with events for estimated upper confidence interval | 3.7 [2.0 to NA] — Insufficient number of participants with events for estimated upper confidence interval | NA [2.1 to NA] — Median duration of PFS not reached; Insufficient number of participants with events for estimated upper confidence interval

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from date of first dose of study treatment to date of death
Time Frame: Up to 31.5 months
Population: Full Analysis Set (FAS) includes all enrolled participants who received any study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A1: CMP-001+Cemiplimab for CSCC | Cohort A2: CMP-001+Cemiplimab for CSCC | Cohort B1: CMP-001+Cemiplimab for MCC | Cohort B2: CMP-001+Cemiplimab for MCC | Cohort D: CMP-001+Cemiplimab for BCC
Number analyzed (Participants) | 25 | 19 | 13 | 16 | 4
Months | 15.6 [10.9 to NA] — Insufficient number of participants with events for estimated upper confidence interval | 12.7 [6.7 to NA] — Insufficient number of participants with events for estimated upper confidence interval | NA [10.9 to NA] — Median duration of PFS not reached; Insufficient number of participants with events for estimated upper confidence interval | 9.9 [4.9 to NA] — Insufficient number of participants with events for estimated upper confidence interval | NA [NA to NA] — Median duration of PFS not reached; Insufficient number of participants with events for estimated lower and upper confidence interval

ADVERSE EVENTS:
Time Frame: From signing of informed consent through end of study up to approximately 31.5 months.
Arm/Group | Cohort A1: CMP-001+Cemiplimab for CSCC | Cohort A2: CMP-001+Cemiplimab for CSCC | Cohort B1: CMP-001+Cemiplimab for MCC | Cohort B2: CMP-001+Cemiplimab for MCC | Cohort D: CMP-001+Cemiplimab for BCC
All-Cause Mortality (participants affected / at risk) | 8/25 | 8/19 | 4/13 | 9/16 | 0/4
Serious Adverse Events (participants affected / at risk) | 14/25 | 11/19 | 6/13 | 11/16 | 2/4
Other Adverse Events (participants affected / at risk) | 24/25 | 19/19 | 13/13 | 15/16 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A1: CMP-001+Cemiplimab for CSCC (N=25) | Cohort A2: CMP-001+Cemiplimab for CSCC (N=19) | Cohort B1: CMP-001+Cemiplimab for MCC (N=13) | Cohort B2: CMP-001+Cemiplimab for MCC (N=16) | Cohort D: CMP-001+Cemiplimab for BCC (N=4)
Injection site reaction (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 3 (3) | 3 (5) | 2 (2) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (5) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral vein stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A1: CMP-001+Cemiplimab for CSCC (N=25) | Cohort A2: CMP-001+Cemiplimab for CSCC (N=19) | Cohort B1: CMP-001+Cemiplimab for MCC (N=13) | Cohort B2: CMP-001+Cemiplimab for MCC (N=16) | Cohort D: CMP-001+Cemiplimab for BCC (N=4)
Fatigue (General disorders) | 15 (29) | 10 (12) | 8 (13) | 8 (16) | 3 (4)
Chills (General disorders) | 10 (19) | 11 (24) | 10 (24) | 8 (13) | 0 (0)
Pyrexia (General disorders) | 6 (9) | 8 (19) | 2 (2) | 4 (6) | 0 (0)
Injection site pain (General disorders) | 4 (4) | 3 (10) | 1 (1) | 2 (2) | 0 (0)
Injection site reaction (General disorders) | 3 (3) | 2 (3) | 0 (0) | 1 (1) | 1 (2)
Oedema peripheral (General disorders) | 3 (4) | 1 (1) | 4 (5) | 3 (3) | 0 (0)
Face oedema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Crepitations (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 2 (11) | 0 (0) | 0 (0)
Obstruction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 3 (8) | 2 (2) | 3 (3) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 9 (12) | 4 (7) | 2 (2) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (9) | 7 (15) | 8 (11) | 5 (6) | 2 (5)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (2) | 2 (2) | 1 (1) | 2 (4)
Constipation (Gastrointestinal disorders) | 4 (5) | 2 (2) | 5 (5) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (10) | 1 (1) | 5 (5) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (3) | 1 (1) | 2 (4) | 2 (3) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 5 (7) | 2 (3) | 3 (4) | 2 (2) | 1 (5)
Alanine aminotransferase increased (Investigations) | 4 (6) | 3 (4) | 3 (4) | 1 (1) | 1 (4)
Lipase increased (Investigations) | 4 (4) | 0 (0) | 2 (3) | 0 (0) | 2 (6)
Lymphocyte count decreased (Investigations) | 4 (5) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 3 (4) | 0 (0) | 2 (3) | 1 (1) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 1 (2)
Weight decreased (Investigations) | 3 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Blood creatinine increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 2 (3) | 0 (0) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Human chorionic gonadotropin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 5 (12) | 5 (7) | 2 (3) | 1 (2)
Dizziness (Nervous system disorders) | 3 (3) | 3 (4) | 3 (3) | 3 (4) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (7) | 4 (6) | 1 (2) | 1 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (5) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 4 (6) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (10) | 3 (4) | 4 (4) | 5 (5) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 4 (6) | 2 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (1) | 4 (15) | 2 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nose deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 2 (3) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 5 (8) | 5 (6) | 1 (2) | 1 (1) | 1 (2)
Hypotension (Vascular disorders) | 4 (12) | 2 (2) | 2 (2) | 4 (9) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 3 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (7) | 1 (2) | 3 (3) | 2 (2) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 2 (4) | 1 (1) | 2 (16) | 0 (0) | 0 (0)
Buttock injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (4) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night blindness (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 2 (2) | 1 (1) | 1 (2) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasm swelling (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (8) | 7 (9) | 1 (1) | 6 (10) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 1 (2) | 2 (3) | 2 (2) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Anhedonia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aural polyp (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Terminated early due to study drug supply. Enrolled 77 of 225 planned participants. Participants only enrolled in CSCC, MCC, & BCC cohorts at time of diagnosis. Results descriptive in nature. No conclusions can be inferred from cohorts analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2023-11-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT04916002/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT04916002/SAP_001.pdf